CLINICAL TRIAL: NCT07124533
Title: Effectiveness of Toothpaste Tablets on Plaque, Gingival Health and Caries Experiences: A 6-week Randomized Controlled Trial
Brief Title: Effectiveness of Toothpaste Tablets on Plaque, Gingival Health and Caries Experiences
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5250357
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gingival Inflammation; Dental Caries
Keywords: Gingival Index; Plaque Index; Dentifrice; Toothpaste Tablets; Caries Experiences; Consumer Satisfaction
MeSH Terms: conditions — Gingivitis; Dental Caries; Consumer Behavior | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Toothpaste Tablet (Experimental): Subjects are instructed to use one toothpaste tablet at each brushing. Brushing is recommended twice daily for two minutes.
  Interventions: Drug: Toothpaste Tablet
- Conventional Toothpaste (Active Comparator): Subjects are instructed to use the toothpaste at each brushing. Brushing is recommended twice daily for two minutes.
  Interventions: Drug: Conventional Toothpaste

INTERVENTIONS:
Drug: Toothpaste Tablet — Denttabs toothpaste tablets
  Other Names: Denttabs Toothpaste Tablets
  Arms: Toothpaste Tablet
Drug: Conventional Toothpaste — Colgate Cavity Protection toothpaste
  Other Names: Colgate Cavity Protection
  Arms: Conventional Toothpaste

SUMMARY:
Objectives: To evaluate the effectiveness of toothpaste tablets when compared to conventional dentifrices in removing plaque.

Methods: 50 participants are randomized into two groups: Denttabs toothpaste tablets (T) and Colgate's Cavity Protection toothpaste (P). Both groups utilize their assigned dentifrice for 6 weeks. A pre and post-assessment measures the Gingival Index (GI) and Plaque Index (PI) and Decayed, Missing and Filled Teeth (DMFT). A questionnaire on the use of the product is distributed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 18 years or older;
2. Subjects who will comply with study protocol;
3. Subjects who can read and understand the consent form;
4. Subjects available during the study period;
5. Subjects have more than 20 teeth.

Exclusion Criteria:

1. Subjects under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Plaque Index Score at Baseline | Change between baseline at visit 1 and visit 2, six weeks post baseline
  The quantity of plaque build-up is measured visually using the Quigley-Hein Plaque Index. The Plaque index can range from 0 to 5, with higher numbers indicating more plaque build-up.
Gingival Index Score at Baseline | Change between baseline at visit 1 and visit 2, six weeks post baseline
  The severity of gingival inflammation is measured visually using the Loe-Silness Gingival Index. Gingival index can range from 0 to 3, with higher numbers indicating more gingival inflammation.

SECONDARY OUTCOMES:
DMFT Score at Baseline | Change between baseline at visit 1 and visit 2, six weeks post baseline
  Caries experiences is measured visually using the DMFT index. DMFT score can range from 0 to 28, with higher numbers indicating higher caries experiences.
Subject Perception of Product Use | Visit 2 six weeks post study enrollment
  The perception on the product usage is measured using a survey containing questions on feel, texture, flavor, ease of use, eco-friendliness, cost and overall satisfaction. Response is on a 4 point Likert scale ranging from strongly agree (1) to strongly disagree (4).

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Kwon, DDS, MS, PhD, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda University Health, Loma Linda, California
  - Loma Linda University, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No